CLINICAL TRIAL: NCT00633022
Title: A Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Effects of Two Regimens of GW856553, Over a Period of 3 Month, on In-vivo Macrophage Activity, as Assessed by FDG-PET/CT Imaging, in the Carotid Arteries and Aorta of Subjects With Established Atherosclerosis
Brief Title: A Study to Evaluate the Effects of 3 Months Dosing With GW856553, as Assessed FDG-PET/CT Imaging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM1111138
Record Dates: First submitted 2008-02-13; First posted 2008-03-11 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis
Keywords: FDG-PET/CT, atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LOSMAPIMOD 7.5 MG TWICE DAILY (Experimental): Participants received 1 tablet of 7.5 mg Losmapimod orally twice daily, each morning and evening for a period of 12 weeks
  Interventions: Drug: LOSMAPIMOD 7.5 MG
- Placebo (Placebo Comparator): Participants received 1 tablet of placebo matching Losmapimod orally twice daily, each morning and evening for a period of 12 weeks.
  Interventions: Drug: Placebo
- LOSMAPIMOD 7.5 MG ONCE DAILY (Experimental): Participants received 1 tablet of 7.5 mg Losmapimod each morning once daily and placebo tablet each evening once daily orally for a period of 12 weeks.
  Interventions: Drug: LOSMAPIMOD 7.5 MG

INTERVENTIONS:
Drug: LOSMAPIMOD 7.5 MG — GW856553 tablets (wet granulation formulation) are available as white, film coated, round, convex tablets manufactured using micronised GW856553X active substance. Tablets are available containing 7.5 mg of GW856553X and are packed into high-density polyethylene (HDPE) bottles.
  Arms: LOSMAPIMOD 7.5 MG ONCE DAILY; LOSMAPIMOD 7.5 MG TWICE DAILY
Drug: Placebo — Placebo tablets (wet granulation formulation) are available as white, film coated, round, convex tablets manufactured using micronised substance to visually match the active GW856553 tablets are also available. Tablets are packed into high-density polyethylene (HDPE) bottles.
  Arms: Placebo

SUMMARY:
This study is being conducted to assess the potential anti-inflammatory effects of a 3-month treatment with GW856553, on the inflammatory activity within the aorta and carotid plaques, as assessed by FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria for Main Study:

1. Adult male and female subjects, between 50 and 80 years of age, inclusive, with a body weight > 50 kg and body mass index (BMI) between 19 and 35 kg/m2
2. Subjects who have:

   * experienced a CV event (acute coronary syndrome, unstable angina, CABG, PCI, stroke, MI, TIA, carotid endarterectomy), but have been clinically stable for at least 6 months since that event,
   * or, have peripheral vascular disease (PVD), as indicated by

     * symptoms of claudication and either a positive imaging/treadmill test, or
     * reduced ankle branchial pressure index,
   * or, have a diagnosis of CAD corroborated by stress testing (exercise or pharmacological) or any other confirmed diagnosis of atherosclerotic arterial disease
   * Individuals who have experienced a CV event or have PVD will be given preference for enrolment in the study, if they also have one of the following:

     * metabolic syndrome, as defined by NCEP ATP III
     * Framingham score > 20
     * Current smokers (at least 1pack/day)
     * Well-controlled diabetes, defined for the purposes of this study as HbA1c <= 8%, or fasting blood glucose <= 126mg/dL (7mmol/L)
3. Subjects must be on a stable dose of statin for at least 3 months prior to first dose of study medication. Subjects must be capable of continuing statin therapy from screening until the final follow up visit.
4. Either carotid or aortic TBR ³ 1.6, as measured on FDG-PET/CT, signifying active inflammation.
5. AST and ALT < 2xULN at screening; alkaline phosphatase and bilirubin <= 1.5xULN at screening (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
6. A signed and dated written informed consent prior to admission to the study
7. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria for Main Study:

1. Any medical history or clinically relevant abnormality identified on the screening medical examination, vital sign measurement, 12-lead ECG recording and/or clinical laboratory examination that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern.
2. History of heart failure defined as NYHA class II - IV or those with known severe LV systolic dysfunction (EF<30%) regardless of symptomatic status
3. Subjects with atrial fibrillation (AF) at screening will be excluded.
4. Insulin controlled Type 1 or Type 2 diabetics
5. Diabetics with fasting glucose > 126mg/dL (7mmol/L) or HbAc1 levels > 8%, at screening. [note: fasting glucose to be checked again at first FDG-PET scan, and if glucose > 11mmol/L at that visit, subject will be excluded from study]
6. Positive pre-study hepatitis B surface antigen or positive hepatitis C antibody results within 3 months of screening.
7. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
8. Renal impairment with creatinine clearance of <40 ml/min at screening, or history of kidney transplant or history of contrast nephropathy.
9. Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with active chronic inflammation (e.g. Inflammatory Bowel Disease).
10. Subjects with chronic infections such as HIV, gingivitis, periodonitis, prostatitis, gastritis, and urinary tract infections, or any active diseases, including active tuberculosis or a history of active tuberculosis.
11. Subjects with any acute infection, symptoms suggestive of sinusitis, or significant trauma (burns, fractures)
12. History of malignancy within the past 5 years, other than non-melanoma skin cancer.
13. History of skeletal muscle myopathy or rhabdomyolysis
14. Previous exposure to GW856553.
15. Current use of steroids (inhaled or oral)
16. Subjects who have donated more than 500 mL of blood within 56 days prior to the study medication administration.
17. Participation in a clinical study where the subject has received a drug or new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of the drug (whichever is longer) prior to the first dose of study medication
18. History of alcohol/drug abuse or dependence within 12 months of the study
19. The subject has a three month prior history of regular alcohol consumption exceeding an average weekly intake of >28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine; or a positive alcohol breath test at the screening visit
20. A positive urine test for drugs of abuse (not related to known medications the subject is taking, e.g. codeine for pain management) or alcohol at screening or prior to study medication administration.
21. QTc interval > 450 msec (using average value of triplicate ECGs)
22. Subjects will be excluded if they have participated in clinical research studies involving radiation in the past three years
23. Women must be of non-childbearing potential [i.e. either postmenopausal or documented hysterectomy - tubal ligation is not sufficient]. For the purposes of this study, post menopausal is defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. Postmenopausal status will be confirmed by serum or urine FSH and oestradiol concentrations at screening, if appropriate. Surgical sterility will be defined as females who have had a hysterectomy and/or bilateral oophorectomy.
24. An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, injectable progesterone, sub-dermal implants or a tubal ligation if the women could become pregnant from the time of the first dose of the study medication until 3 months after administration of last dose of study medication.

Inclusion Criteria for Subjects in MRI Sub-study

1. Recent (in approximately last 12 months) echocardiogram with ejection fraction between 30 and 50%.

Exclusion Criteria for Subjects in MRI Sub-study

1. Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but not limited to:

   * Intracranial aneurysm clips (except Sugita) or other metallic objects,
   * History of intra- orbital metal fragments that have not been removed by an MD,
   * Pacemakers, implantable cardiac defibrillators and non-MR compatible heart valves,
   * Inner ear implants,
   * History of claustrophobia in MR.
2. Allergy to MRI contrast enhancement agent (gadolinium).
3. Serum creatinine clearance < 60 mL/min (At the discretion of the physician, the subject may progress to a formal assessment based on 24 hour urine collection should serum creatinine limits fall below limits.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-06-02 (Actual); Primary Completion 2009-12-03 (Actual); Study Completion 2009-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Elkhawad M, Rudd JH, Sarov-Blat L, Cai G, Wells R, Davies LC, Collier DJ, Marber MS, Choudhury RP, Fayad ZA, Tawakol A, Gleeson FV, Lepore JJ, Davis B, Willette RN, Wilkinson IB, Sprecher DL, Cheriyan J. Effects of p38 mitogen-activated protein kinase inhibition on vascular and systemic inflammation in patients with atherosclerosis. JACC Cardiovasc Imaging. 2012 Sep;5(9):911-22. doi: 10.1016/j.jcmg.2012.02.016. PMID 22974804
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: PM1111138 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with established atherosclerosis were planned to be enrolled across 4 sites in the United Kingdom from 02 June 2008 to 03 December 2009. Participants were screened within 45 days prior to the first dose and underwent radiological scan within 14 days prior to the first dose.
Pre-assignment Details: Participants were randomized in the study to receive oral dose of Losmapimod 7.5 milligram (mg) twice daily, Losmapimod 7.5 mg once daily or placebo.
Period: Overall Study
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Started | 34 | 33 | 32
Completed | 33 | 32 | 27
Not Completed | 1 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 5
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo | Total
Number analyzed (Participants) | 34 | 33 | 32 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (5.90) | 65.3 (5.94) | 63.7 (6.37) | 63.8 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 14
  Male | 29 | 28 | 28 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 32 | 30 | 30 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Mean of Maximum Tissue to Background Ratio (TBR) in the Qualifying Artery, Following 12 Weeks of Treatment in the Setting of Chronic Statin Therapy
Description: Qualifying artery was defined as the artery (left or right carotid or ascending aorta) with the highest segmental mean of maximum (max) TBR at Baseline. The TBR of the qualifying segment was to be ≥ 1.6. If more than one artery qualified, the hottest (greatest mean of max TBR) artery was the qualifying artery. Baseline was defined as the value between Days -14 to -1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-treatment values.
Time Frame: Baseline (Days -14 to -1) and up to Week 12
Population: Pharmacodynamic (PD) Population comprised of all participants who provided PD data. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Maximum tissue to background ratio
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 32 | 32 | 29
Maximum tissue to background ratio | -0.146 (0.2483) | -0.122 (0.1839) | -0.070 (0.1632)
Statistical Analysis 1: Comparison: Losmapimod 7.5 mg Twice Daily vs Placebo; Losmapimod 7.5 mg BID versus Placebo; Test type: Superiority; p = 0.4519, ANCOVA; ANCOVA model, fitting fixed effect treatment term, and including baseline TBR value as a covariate.ANCOVA model, fitting fixed effect treatment term,; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.14 to 0.06] — The point estimate was calculated as least square mean difference (final values) of Losmapimod 7.5 mg twice daily and Placebo
Statistical Analysis 2: Comparison: Losmapimod 7.5 mg Once Daily vs Placebo; Losmapimod 7.5 mg once daily versus Placebo; Test type: Superiority; p = 0.5789, ANCOVA; ANCOVA model, fitting fixed effect treatment term, and including baseline TBR value as a covariate; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.11 to 0.06] — The point estimate was calculated as least square mean difference (final values) of Losmapimod 7.5 mg once daily and Placebo

2. Secondary Outcome: Change From Baseline of the 'Most Diseased Segment (MSD)' Average Maximum TBR in the Qualifying Artery Following 12 Weeks of Treatment With GW856553 or Placebo in the Setting of Chronic Statin Therapy
Description: Most diseased segment (MDS) mean of max TBR was mean of all the slice max TBR that compose the most diseased segment. TBR was derived by dividing the arterial vessel wall SUV (tissue) by the background venous blood pool SUV. Unless noted otherwise, the tissue max SUV value for each ROI was used as inputs to the TBR. Baseline was defined as the value between Days -14 to -1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-treatment values.
Time Frame: Baseline (Days -14 to -1) and up to Week 12
Population: PD Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 31 | 32 | 28
Ratio | -0.294 (0.3169) | -0.250 (0.2892) | -0.221 (0.2132)
Statistical Analysis 1: Comparison: Losmapimod 7.5 mg Twice Daily vs Placebo; Losmapimod 7.5 mg twice daily versus placebo; Test type: Superiority; p = 0.6986, ANCOVA; ANCOVA model, fitting fixed effect treatment term, and including baseline TBR value as a covariate; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.15 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Losmapimod 7.5 mg Once Daily vs Placebo; Losmapimod 7.5 mg once daily versus Placebo; Test type: Superiority; p = 0.9486, ANCOVA; ANCOVA model, fitting fixed effect treatment term, and including baseline TBR value as a covariate; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.13 to 0.12] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline in Blood Concentration of High Sensitivity C-reactive Protein (Hs-CRP)
Description: CRP is a protein that the liver makes when there is inflammation in the body. It's also called a marker of inflammation, and can be measured with an hs-CRP test. Blood samples were collected to analyze hs-CRP. Baseline was defined as the value on Day 1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-treatment values.
Time Frame: Baseline (Day 1) and Days 7, 14, 21, 28, 42, 56, 70, 84
Population: PD Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: milligram per litre (mg/L)
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
milligram per litre (mg/L)
  Day 7: number analyzed (Participants) | 15 | 13 | 14
  Day 7 | -2.293 (6.0389) | -0.446 (0.5547) | 0.079 (0.6886)
  Day 14: number analyzed (Participants) | 32 | 30 | 31
  Day 14 | -0.756 (4.8068) | -0.617 (2.0800) | -0.352 (1.9871)
  Day 21: number analyzed (Participants) | 14 | 10 | 12
  Day 21 | -2.250 (5.9883) | 0.130 (1.1586) | 0.242 (1.3125)
  Day 28: number analyzed (Participants) | 31 | 30 | 31
  Day 28 | -1.394 (3.9276) | 1.953 (13.6807) | 0.197 (3.7474)
  Day 42: number analyzed (Participants) | 13 | 11 | 11
  Day 42 | -0.085 (10.3631) | -0.145 (0.6186) | -0.009 (0.8105)
  Day 56: number analyzed (Participants) | 32 | 30 | 27
  Day 56 | 0.012 (6.0287) | 0.077 (4.6724) | 0.563 (5.0270)
  Day 70: number analyzed (Participants) | 8 | 7 | 7
  Day 70 | 1.313 (2.8216) | 0.086 (0.9118) | -0.657 (1.3011)
  Day 84: number analyzed (Participants) | 29 | 29 | 24
  Day 84 | -0.100 (1.5281) | 1.452 (5.3392) | -0.313 (1.9369)

4. Secondary Outcome: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points
Description: Blood pressure measurements were taken to observe vital signs and included SBP and DBP. SBP and DBP measurements were obtained at Day 1, 7, 14, 21, 28, 42, 56, 70, 84 and follow-up (1-2 weeks post last dose on Day 84).
Time Frame: Day 1, 7, 14, 21, 28, 42, 56, 70, 84, 98
Population: Safety Population comprised of all participants who received at least one dose of study drug. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mm/Hg)
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
millimeter of mercury (mm/Hg)
  DBP: Day 1 | 78.9 (8.67) | 76.7 (11.08) | 75.8 (7.64)
  DBP: Day 7: number analyzed (Participants) | 16 | 15 | 14
  DBP: Day 7 | 79.4 (8.00) | 73.6 (11.04) | 73.9 (6.81)
  DBP: Day 14: number analyzed (Participants) | 34 | 32 | 32
  DBP: Day 14 | 76.6 (9.01) | 76.1 (10.55) | 76.4 (9.03)
  DBP: Day 21: number analyzed (Participants) | 15 | 12 | 13
  DBP: Day 21 | 77.9 (8.44) | 73.8 (12.05) | 74.5 (7.60)
  DBP: Day 28 | 77.4 (9.64) | 76.5 (9.63) | 76.4 (8.96)
  DBP: Day 42: number analyzed (Participants) | 13 | 12 | 11
  DBP: Day 42 | 80.6 (11.12) | 72.8 (8.96) | 74.6 (7.94)
  DBP: Day 56: number analyzed (Participants) | 34 | 32 | 29
  DBP: Day 56 | 77.5 (10.95) | 75.7 (9.09) | 75.9 (7.50)
  DBP: Day 70: number analyzed (Participants) | 7 | 8 | 7
  DBP: Day 70 | 76.3 (4.54) | 73.8 (10.71) | 75.0 (6.30)
  DBP: Day 84: number analyzed (Participants) | 32 | 30 | 26
  DBP: Day 84 | 75.6 (8.68) | 75.4 (9.51) | 76.2 (8.90)
  DBP: Day 98: number analyzed (Participants) | 34 | 33 | 31
  DBP: Day 98 | 78.0 (9.81) | 76.6 (10.58) | 73.6 (8.26)
  SBP: Day 1 | 134.9 (16.67) | 132.6 (16.00) | 129.5 (19.22)
  SBP: Day 7: number analyzed (Participants) | 16 | 15 | 14
  SBP: Day 7 | 132.4 (19.40) | 123.1 (13.58) | 122.4 (13.99)
  SBP: Day 14: number analyzed (Participants) | 34 | 32 | 32
  SBP: Day 14 | 128.2 (17.08) | 133.3 (19.05) | 130.3 (17.87)
  SBP: Day 21: number analyzed (Participants) | 15 | 12 | 13
  SBP: Day 21 | 136.9 (15.12) | 132.8 (20.80) | 126.6 (15.76)
  SBP: Day 28 | 131.7 (21.94) | 132.3 (17.79) | 128.5 (18.76)
  SBP: Day 42: number analyzed (Participants) | 13 | 12 | 11
  SBP: Day 42 | 140.7 (19.78) | 126.5 (17.94) | 128.3 (20.10)
  SBP: Day 56: number analyzed (Participants) | 34 | 32 | 29
  SBP: Day 56 | 130.1 (17.88) | 130.5 (16.91) | 127.4 (16.69)
  SBP: Day 70: number analyzed (Participants) | 7 | 8 | 7
  SBP: Day 70 | 136.3 (11.46) | 122.8 (14.56) | 135.4 (19.48)
  SBP: Day 84: number analyzed (Participants) | 32 | 30 | 26
  SBP: Day 84 | 129.5 (17.78) | 128.1 (14.32) | 126.4 (19.84)
  SBP: Day 98: number analyzed (Participants) | 34 | 33 | 31
  SBP: Day 98 | 131.2 (18.06) | 130.9 (17.61) | 125.1 (15.87)

5. Secondary Outcome: Mean Heart Rate at Indicated Time Points
Description: Vital sign monitoring included heart rate measurement. Heart rate measurements were obtained at Day 1, 7, 14, 21, 28, 42, 56, 70, 84 and follow-up (1-2 weeks post last dose on Day 84).
Time Frame: Day 1, 7, 14, 21, 28, 42, 56, 70, 84, 98
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
beats per minute (bpm)
  Heart rate: Day 1 | 57.6 (11.39) | 56.3 (9.84) | 56.5 (9.79)
  Heart rate: Day 7: number analyzed (Participants) | 16 | 15 | 14
  Heart rate: Day 7 | 60.8 (13.97) | 52.5 (6.81) | 54.6 (6.11)
  Heart rate: Day 14: number analyzed (Participants) | 34 | 32 | 32
  Heart rate: Day 14 | 57.7 (11.80) | 56.7 (7.66) | 55.4 (10.32)
  Heart rate: Day 21: number analyzed (Participants) | 15 | 12 | 13
  Heart rate: Day 21 | 63.9 (12.44) | 54.3 (6.59) | 54.8 (8.97)
  Heart rate: Day 28: number analyzed (Participants) | 34 | 32 | 32
  Heart rate: Day 28 | 58.7 (12.25) | 56.4 (9.17) | 57.2 (10.91)
  Heart rate: Day 42: number analyzed (Participants) | 13 | 12 | 11
  Heart rate: Day 42 | 60.1 (9.31) | 52.1 (6.46) | 56.8 (10.80)
  Heart rate: Day 56: number analyzed (Participants) | 34 | 32 | 29
  Heart rate: Day 56 | 58.6 (11.48) | 56.1 (10.12) | 56.5 (10.73)
  Heart rate: Day 70: number analyzed (Participants) | 7 | 8 | 7
  Heart rate: Day 70 | 57.3 (7.67) | 53.8 (5.26) | 54.3 (9.52)
  Heart rate: Day 84: number analyzed (Participants) | 32 | 30 | 26
  Heart rate: Day 84 | 58.7 (12.07) | 59.2 (10.35) | 55.8 (11.53)
  Heart rate: Day 98: number analyzed (Participants) | 34 | 33 | 31
  Heart rate: Day 98 | 61.5 (12.09) | 58.2 (9.00) | 56.1 (9.76)

6. Secondary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Findings
Description: All 12-lead ECGs were obtained after the participant had rested in the supine position for at least 15 minutes. All ECGs were evaluated by the principal investigator or designee for any other abnormality of potential clinical importance (PCI). Data for abnormal ECG findings have been reported under abnormal - Not clinically significant (NCS) and Abnormal - Clinically significant (CS) categories. Data only for categories with values have been presented.
Time Frame: Days 1, 7, 14, 21, 28, 42, 56, 70, 84, 98
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Participants
  Day 1 pre-dose 1: Abnormal-NCS | 19 | 17 | 15
  Day 1 pre-dose 2:Abnormal-NCS | 19 | 16 | 15
  Day 1 pre-dose 3: Abnormal-NCS | 18 | 16 | 15
  Day 7 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 16 | 15 | 15
  Day 7 pre-dose 1: Abnormal-NCS | 8 | 8 | 7
  Day 14 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 34 | 32 | 32
  Day 14 pre-dose 1: Abnormal-NCS | 16 | 17 | 16
  Day 28 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 34 | 32 | 32
  Day 28 pre-dose 1: Abnormal-NCS | 16 | 14 | 13
  Day 28 pre-dose 1: Abnormal-CS: number analyzed (Participants) | 34 | 32 | 32
  Day 28 pre-dose 1: Abnormal-CS | 0 | 0 | 1
  Day 56 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 34 | 32 | 29
  Day 56 pre-dose 1: Abnormal-NCS | 17 | 15 | 12
  Day 70 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 7 | 8 | 7
  Day 70 pre-dose 1: Abnormal-NCS | 4 | 4 | 4
  Day 84 pre-dose 1: Abnormal-NCS: number analyzed (Participants) | 33 | 32 | 27
  Day 84 pre-dose 1: Abnormal-NCS | 15 | 17 | 11
  Day 98: Abnormal-NCS: number analyzed (Participants) | 34 | 33 | 31
  Day 98: Abnormal-NCS | 15 | 18 | 13
  Day 98: Abnormal-CS: number analyzed (Participants) | 34 | 33 | 31
  Day 98: Abnormal-CS | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Clinical Chemistry Abnormalities of PCI
Description: Clinical chemistry range for PCI was calcium low <1.5 mill mole per litre (mmol/L), high > 3.24 mmol/L; creatinine high 155 mmol/L; glucose low < 2.2 (age: 13-99) mmol/L, high > 27.8 (age: 13-99) mmol/L; phosphorus low < 2.8 mmol/L, high > 6.5 mmol/L; sodium low < 125 mmol/L, high > 150 mmol/L. Categories with values have been presented.
Time Frame: Up to Follow-up (Day 98)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Participants
  Calcium low | 2 | 0 | 0
  Calcium high | 0 | 0 | 1
  Glucose low | 1 | 0 | 0
  Glucose high | 7 | 2 | 3
  Potassium low | 1 | 2 | 0
  Sodium low | 1 | 3 | 3
  Creatinine high | 0 | 2 | 4
  Chloride low | 0 | 2 | 0

8. Secondary Outcome: Number of Participants With Hematology Abnormalities of PCI
Description: Hematology range for PCI was: white blood cell count (WBC) low < 1.1 x109/ L; hemoglobin low <71 (age: 18-99) grams per litre (g/L), high >199 (age: 18-99) g/L; hematocrit low 0.201 (age: 18-99) ratio of 1 high 0.599 (age: 18-99) ratio of 1 and platelet count low < 80 x109/ L, high > 500 x109/ L. Categories with values have been presented.
Time Frame: Up to Follow-up (Day 98)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Participants
  Eosinophils high | 3 | 1 | 1
  Eosinophils low | 0 | 0 | 1
  Haemoglobin low | 1 | 0 | 1
  Lymphocytes low | 4 | 2 | 2
  Lymphocytes high | 1 | 0 | 2
  MCH high | 0 | 0 | 1
  Monocytes high | 1 | 0 | 1
  Neutrophils low | 0 | 0 | 1
  Neutrophils high | 3 | 1 | 0
  RBC count low | 1 | 0 | 1
  Reticulocytes low | 4 | 4 | 9
  Reticulocytes high | 18 | 10 | 13
  Platelet count low | 0 | 1 | 0
  WBC count low | 0 | 1 | 0

9. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results
Description: A urine dipstick test is a basic diagnostic tool used to determine pathological changes in a participant's urine in standard urinalysis. Data was analyzed for urine occult blood, urine glucose, urine ketones and urine protein ranging from 2+, trace, 1+, 3+, 1+or 1/4, 3+ or 1 and trace or 1/10, indicating proportional concentrations in the urine sample. Data has been presented for categories with values for positive findings.
Time Frame: Day 1, 7, 14, 21, 28, 42, 56, 70, 84, 98
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Participants
  Day 1: Urine Occult Blood, trace | 1 | 1 | 2
  Day 1: Urine Occult Blood, 3+ | 0 | 0 | 1
  Day 1: Urine Glucose, 1+ | 0 | 0 | 1
  Day 1: Urine Protein, trace | 4 | 1 | 2
  Day 1: Urine Protein, 1+ | 2 | 0 | 5
  Day 7: Urine Occult Blood, 1+ | 0 | 0 | 1
  Day 7: Urine Occult Blood, 3+ | 0 | 0 | 1
  Day 7: Urine Protein, trace | 0 | 1 | 3
  Day 7: Urine Protein, 1+ | 1 | 0 | 1
  Day 14: Urine Occult Blood, 2+ | 0 | 0 | 1
  Day 14: Urine Occult Blood, trace | 1 | 2 | 0
  Day 14: Urine Occult Blood, 1+ | 0 | 0 | 3
  Day 14: Urine Ketones, trace | 0 | 1 | 0
  Day 14: Urine Protein, trace | 1 | 1 | 3
  Day 14: Urine Protein, 1+ | 3 | 0 | 2
  Day 21: Urine Occult Blood, trace | 1 | 0 | 0
  Day 21: Urine Ketones, trace | 0 | 0 | 1
  Day 21: Urine Protein, trace | 1 | 0 | 3
  Day 21: Urine Protein, 1+ | 1 | 0 | 1
  Day 28: Urine Occult Blood, 2+ | 0 | 0 | 2
  Day 28: Urine Occult Blood, trace | 1 | 1 | 1
  Day 28: Urine Protein, trace | 2 | 3 | 5
  Day 28: Urine Protein, 1+ | 3 | 0 | 1
  Day 42: Urine Occult Blood, 2+ | 0 | 0 | 1
  Day 42: Urine Protein, trace | 0 | 1 | 2
  Day 42: Urine Protein, 1+ | 1 | 0 | 0
  Day 56: Urine Occult Blood, 2+ | 0 | 0 | 1
  Day 56: Urine Occult Blood, trace | 0 | 0 | 2
  Day 56: Urine Occult Blood, 1+ | 0 | 1 | 2
  Day 56: Urine Glucose, Trace or 1/10 | 0 | 0 | 1
  Day 56: Urine Ketones, trace | 1 | 0 | 0
  Day 56: Urine Protein, trace | 2 | 2 | 1
  Day 56: Urine Protein, 1+ | 3 | 0 | 2
  Day 70: Urine Occult Blood, 2+ | 0 | 0 | 1
  Day 70: Urine Occult Blood, trace | 1 | 0 | 0
  Day 70: Urine Protein, 2+ | 1 | 0 | 0
  Day 70: Urine Protein, trace | 0 | 0 | 1
  Day 70: Urine Protein, 1+ | 0 | 0 | 1
  Day 84: Urine Occult Blood, 2+ | 0 | 1 | 1
  Day 84: Urine Occult Blood, trace | 0 | 0 | 1
  Day 84: Urine Occult Blood, 1+ | 0 | 0 | 2
  Day 84: Urine Ketones, trace | 0 | 0 | 1
  Day 84: Urine Protein, 2+ | 0 | 1 | 0
  Day 84: Urine Protein, trace | 2 | 3 | 5
  Day 84: Urine Protein, 1+ | 3 | 0 | 0
  Day 98: Urine Occult Blood, 2+ | 0 | 0 | 1
  Day 98: Urine Occult Blood, trace | 1 | 1 | 0
  Day 98: Urine Occult Blood, 1+ | 0 | 1 | 1
  Day 98: Urine Occult Blood, 3+ | 0 | 0 | 1
  Day 98: Urine Glucose, 3+ OR 1 | 0 | 1 | 0
  Day 98: Urine Protein, trace | 2 | 1 | 3
  Day 98: Urine Protein, 1+ | 3 | 0 | 3

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Follow-up (Day 98)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Participants
  Any AE | 29 | 28 | 31
  Any SAE | 4 | 1 | 3

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected up to Follow-up visit (Day 98)
Description: SAEs and non-serious AEs are reported for Safety Population.
Arm/Group | Losmapimod 7.5 mg Twice Daily | Losmapimod 7.5 mg Once Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 1/32
Serious Adverse Events (participants affected / at risk) | 4/34 | 1/33 | 3/32
Other Adverse Events (participants affected / at risk) | 25/34 | 24/33 | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 7.5 mg Twice Daily (N=34) | Losmapimod 7.5 mg Once Daily (N=33) | Placebo (N=32)
Meningitis herpes (Infections and infestations) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Road trafic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 7.5 mg Twice Daily (N=34) | Losmapimod 7.5 mg Once Daily (N=33) | Placebo (N=32)
Headache (Nervous system disorders) | 7 | 10 | 10
Dizziness (Nervous system disorders) | 2 | 2 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 4
Migraine (Nervous system disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1
Toothache (Gastrointestinal disorders) | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 5
Chest pain (General disorders) | 3 | 2 | 2
Chest discomfort (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Palpitations (Cardiac disorders) | 2 | 3 | 1
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 3 | 0
Blood urine present (Investigations) | 0 | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Eye pain (Eye disorders) | 0 | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0
Depressed mood (Psychiatric disorders) | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Tooth extraction (Surgical and medical procedures) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.